CLINICAL TRIAL: NCT00298883
Title: Desensitization of Renal Transplant Candidates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 584-2004
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: End Stage Renal Disease; Kidney Transplantation
Keywords: Renal; Transplant; PRA
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): This is a single arm, interventional trial.
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — Myfortic 360mg PO BID for six weeks

SUMMARY:
Trial of the use of Myfortic to reduce anti-HLA alloantibody in patients waiting for renal transplantation.

DETAILED DESCRIPTION:
Pre-formed HLA antibodies prevent renal transplantation because of the risk of hyperacute rejection. We propose a prospective study evaluating the efficacy of Enteric Coated Mycophenolate Sodium (Myfortic) in decreasing the titers of anti-HLA alloantibodies in patients awaiting kidney transplantation. Myfortic is an immunosuppressant that inhibits the proliferation of B and T cells by blocking the enzyme inosine monophosphate dehydrogenase. We will attempt to determine whether a 6-week course of Myfortic adequately decreases the antibody reactivity to a level compatible with transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the deceased donor kidney transplant waiting list with panel reactive antibodies >50% and living donor waiting list patients who have a history of a positive crossmatch (donor-specific antibodies) will be eligible for the study.

Exclusion Criteria:

* Any subjects not meeting the Inclusion Criteria
* Subjects unable to attend weekly clinic visits for six weeks
* Inability to tolerate Myfortic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
decrease in antibody reactivity | six weeks

SECONDARY OUTCOMES:
CBC and CMP values </> 2 times normal | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shiro Fujita, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States